CLINICAL TRIAL: NCT04813068
Title: A Qualitative Study of Patients' Attitudes to the Risks and Potential Benefits of Potential Toxicities of Radical Re-irradiation for Lung Cancer
Brief Title: Lung Cancer Patients' Attitudes to a Second Course of Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); The Beatson Cancer Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: GN20ON632
Record Dates: First submitted 2021-03-12; First posted 2021-03-24 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer; Recurrence
MeSH Terms: conditions — Lung Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview arm: Group of patients who have agreed to have a qualitative interview on the topic of recurrence of lung cancer
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interview to identify attitudes to re-irradiation in lung cancer

SUMMARY:
Patients with lung cancer are often treated with high dose x-ray treatment (radical radiotherapy) to control the disease. After one course of radiotherapy, after a period of time, there is a risk that the cancer can come back in either the same place or nearby in the lungs. This happens to about 700 patients in the UK every year. There is no strong evidence to suggest what the best treatment is in this situation.

One possible treatment is a second course of radiotherapy (re-irradiation). Early studies show that a re-irradiation may cause significant side effects like breathlessness or problems swallowing, but may control the cancer for a long period of time. We want to do a clinical trial to investigate if re-irradiation improves cancer control compared to other treatments to help guide treatment for patients with recurrent disease.

Before we can go ahead with the trial, we would like to talk to patients who are have completed radiotherapy to find out what are their feelings about having a second course of radiotherapy if needed, and how the side effects from the initial course of radiotherapy or the projected side-effects from the second course would affect that decision.

This information is vitally important to help develop a trial about re-irradiation in lung cancer as it will demonstrate if patients would accept a second course of radiotherapy, and, by accounting for patient concerns in the trial design, will make it more likely to recruit well.

This study will perform telephone interviews with patients five weeks after completing a course of radical radiotherapy for lung cancer at the Beatson Cancer Centre. We expect to interview 16-30 patients. This study will run over the course of 1 year. This research is funded by the Beatson Cancer Charity and The University of Glasgow.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Pathological or radiological diagnosis of non-small cell lung cancer
* Undergoing radical radiotherapy to the thorax using the following fractionations (55 Gray in 20 fractions, 54 Gray in 36 fractions or any Stereotactic Ablative Body Radiotherapy (SABR) fractionation that delivers a biological effective dose of greater than 100Gy10) as part of their primary lung cancer treatment at time of study enrolment
* Patients receiving concurrent and/or adjuvant systemic therapies are permitted
* Radiotherapy is delivered in the Beatson West of Scotland Cancer Centre
* Signed, written informed consent
* Willing and able to complete study processes

Exclusion Criteria:

* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are having radical radiotherapy for non-small cell lung cancer in the Beatson West of Scotland Cancer Centre, who are consent to a semi-structured interview about their experience of radiotherapy and their feelings on re-treatment if necessary
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Feelings and concerns re: second radiotherapy course | Dec 2021
  Explore patients' feelings and concerns about having a second course of radiotherapy for recurrent lung cancer. This will be assessed using thematic analysis of the transcripts of semi-structured interviews, and the outcome will be the identification of themes that participants have expressed with regard to a second course of radiotherapy e.g. "side-effects of radiotherapy", or "cost of another treatment".

SECONDARY OUTCOMES:
Choice of treatment in recurrent setting | Dec 2021
  Identify factors that patients consider when deciding on potential treatments in the setting of locally recurrent lung cancer (including effect of COVID-19 on treatment choice). This will be assessed using thematic analysis of the transcripts of semi-structured interviews, and the outcome will be the identification of themes that participants have expressed with regard to a choosing a treatment in the event of relapse e.g. "worry about chemotherapy side-effects", or "risk of infection".
Attitude to side effects in context of possible outcomes | Dec 2021
  Investigate how patients' acceptance of side effects changes with the different projected outcomes of re-irradiation. This will be assessed using thematic analysis of the transcripts of semi-structured interviews, and the outcome will be the identification of any hierarchy of side-effects that patients would rather not experience e.g. "I can cope with fatigue but I don't want to be breathless".
Toxicity from previous radiotherapy | Dec 2021
  Explore the relationship between the toxicities patients experienced during radiotherapy and their attitudes to a second course of radiotherapy. As part of the semi-structured interview, participants will be asked to grade the severity of symptoms on a three point scale (mild/moderate/severe) and then state if they would consider a second course of radiotherapy if needed (yes/no). There will be scope in the semi-structured interview to expand on any topic, and this will undergo thematic analysis.
Attitude to surveillance scans | Dec 2021
  Investigate patients' awareness of surveillance imaging after radical treatment and willingness for scans. This will be assessed using thematic analysis of the transcripts of semi-structured interviews, and the outcome will be the identification of themes that participants have expressed with regard to a surveillance e.g. "I'd prefer to have frequent scans to see if there is any change in the tumour", or "frequent scans make me anxious".

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrow, PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- The Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Transcribed and anonymised interviews will be available on the University of Glasgow research repository after the trial has completed

DOCUMENTS (1):
  • Study Protocol (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04813068/Prot_000.pdf